CLINICAL TRIAL: NCT04393220
Title: Combination of PD-1 and VEGFR-2 Blockade for Advanced Hepatocellular Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fuda Cancer Hospital, Guangzhou (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML-20200511
Record Dates: First submitted 2020-05-11; First posted 2020-05-19 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2020-06

CONDITIONS: Progress Free Survival (PFS) and Overall Survival (OS)
MeSH Terms: interventions — Bevacizumab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bevacizumab and anti-PD-1 therapy (Experimental)
  Interventions: Drug: Bevacizumab Injection; Drug: Nivolumab
- Bevacizumab (Active Comparator)
  Interventions: Drug: Bevacizumab Injection
- anti-PD-1 (Active Comparator)
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Bevacizumab Injection — 15mg/kg (Q3W)
  Arms: Bevacizumab; Bevacizumab and anti-PD-1 therapy
Drug: Nivolumab — nivolumab 480 mg IV infusions for 30 minutes q4w
  Arms: Bevacizumab and anti-PD-1 therapy; anti-PD-1

SUMMARY:
The aie of this clinical study is the safety and efficacy of combination therapy for HCC patients.

DETAILED DESCRIPTION:
Activation of anti-tumor immune response using programmed death receptor-1 (PD-1)blockade showed benefit only in a fraction of hepatocellular carcinoma (HCC) patients. Specific blockade of vascular endothelial receptor 2 (VEGFR-2) using a murine antibody significantly delayed primary tumor growth but failed to prolong survival. Combining PD-1 blockade with antiangiogenesis has shown promise in substantially increasing the fraction of HCC patients who respond to treatment in vitro. Based on these clinical data, we are aimed to investigation the safety and efficacy of combination therapy for HCC patients.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 18-70 (inclusive), male and female

  2. HCC was diagnosed by histopathological examination or the guidelines for the diagnosis and treatment of primary liver cancer (2017 edition).

  3. Stage B (intermediate) or stage C (advanced) HCC was determined according to the Barcelona clinical liver cancer staging (BCLC stage).If it is stage B, the patient must be ineligible for surgery and/or local treatment, or develop disease following surgery and/or local treatment, or the patient rejects surgery and/or local treatment (must be specified and signed).

  4. I have not received any systemic therapy for HCC (mainly including systemic chemotherapy, anti-vascular therapy, molecular targeted therapy and immunotherapy containing ctla-4, pd-1 / pd-l1 monoclonal antibody).

  5. according to RECISTv1.1 criteria, there were ≥ 1 measurable lesion.Requirements: the selected target lesion had not received local treatment before, or the selected target lesion was located in the previously treated area, and was later confirmed as PD by imaging examination.

  6. child-pugh liver function grade A, and no history of hepatic encephalopathy. 7. The ECOG (tumor cooperative group in the eastern United States) physical status score (PS) was 0 to 1.

  8. expected survival ≥12 weeks.

  9. Major organ functions meet the following requirements: no blood transfusion, no use of hematopoietic stimulators (including g-csf, gm-csf, EPO and TPO) and infusion of human albumin preparations within 14 days prior to screening: neutrophil absolute count ≥1.5×109/L;Platelet count ≥ 80×109/L;Hemoglobin ≥ 90 g/L;Serum albumin ≥ 29 g/L;Total serum bilirubin ≤1.5× upper limit of normal range (ULN);Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 5 × ULN;Serum creatinine (Cr) ≤1.5×ULN or Cr clearance ≥40 mL/min (calculated by Cockcroft-Gault formula);International standardized ratio (INR) ≤2 or prothrombin time (PT) exceeding the upper limit of normal range ≤6 seconds;Urine protein & lt;2+ (if urine protein ≥2+, 24-hour (h) urine protein quantification and 24h urine protein quantification should be performed <1.0g can be enrolled).

  10. if HBsAg(+) and/or HBcAb(+) are required, HBV DNA must <500IU/mL (if the lower limit of the minimum detectable value of the local center is higher than 500IU/mL, after discussion with the sponsor, the enrollment can be decided according to the specific situation), and the patients should continue to receive the effective anti-hbv treatment that has been adopted or start to use entecavir or tenofovir throughout the study period. Co-infection with HBV and HCV was excluded. Patients with a history of HCV infection but negative PCR results for HCV RNA may be considered to be free of HCV infection.

  11. Women of childbearing age must undergo a blood pregnancy test within the first 7 days of randomization with negative results and agree to use a reliable and effective method of contraception during the trial and within 60 days of the last trial drug administration. Male patients whose partners are women of childbearing age must agree to use a reliable and effective method of contraception during the trial and within 60 days of the last trial drug administration.

  12. Patients voluntarily participated, fully informed consent, and signed written informed consent, with good compliance.

Exclusion Criteria:

* 1. known as cholangiocarcinoma (ICC) or mixed hepatocellular carcinoma, sarcomatoid hepatocellular carcinoma, and hepatic fibrolamellar carcinoma.

  2. Had developed malignant tumor other than HCC within 2 to 5 years;However, limited tumors treated by the study were excluded, including carcinoma in situ of the cervix, basal cell carcinoma of the skin, and carcinoma in situ of the prostate.

  3. had undergone liver surgery and/or local or experimental drug therapy for HCC in the first 4 weeks of randomization;Palliative radiotherapy for bone metastases was performed in the first 2 weeks of randomization.The toxic reaction (except hair loss) caused by previous treatment did not recover to ≤1 (nci-ctc AE v 5.0).Within 2 weeks prior to randomization, a Chinese medicine preparation with anti-hepatocellular carcinoma effect was received.

  4. screening is not the control of pericardial effusion, uncontrolled pleural effusion or clinically significant moderate peritoneal effusion, defined as to the following criteria: screening, have clinical symptom and physical examination can detect the thoracic and abdominal cavity effusion or in the process of screening, need for thoracic and abdominal cavity effusion puncture pumping cavities or fluid and medication.

  5. A history of gastrointestinal bleeding in the first 6 months;In patients with portal hypertension, the researchers concluded that patients with a high risk of bleeding (including moderate to severe esophageal and gastric varices at risk of bleeding, locally active gastrointestinal ulcers, and persistent positive fecal occult blood) should undergo gastroscopy to exclude patients with "red sign".If there is a "red sign" in the history of gastroscopy, it should be excluded from the group.

  6. Present with grade ≥3 (nci-tc AE v5.0) gastrointestinal or non-gastrointestinal fistula.

  7. The main portal vein tumor thrombus (Vp4) or inferior vena cava tumor thrombus should be excluded.However, patients with a main portal vein tumor thrombus but unobstructed branches of the contralateral portal vein may be admitted.

  8. Previous history of serious cardiovascular and cerebrovascular diseases: congestive heart failure, unstable angina, myocardial infarction or cerebrovascular accident stroke of New York cardiology association (NYHA) level II or above occurred in the 12 months before enrollment, or poorly controlled arrhythmias.Cardiac ultrasound examination of LVEF (left ventricular ejection fraction) <50%.Corrected QT interval (QTc) >480ms (calculated using the Fridericia method, if QTc is abnormal, it can be detected for 3 times at an interval of 2 minutes, and the average value is taken).High blood pressure (systolic blood pressure (BP) ≥150 mmHg and/or diastolic blood pressure ≥100mmHg) (mean of ≥3 BP readings based on ≥2 measurements) that are difficult to control with medication.Hypertensive crisis or hypertensive encephalopathy occurred in the past.

  9. Significant bleeding disorder or other evidence of significant bleeding tendency: clinically significant hemoptysis or tumor bleeding of any cause occurred within 2 weeks prior to enrollment;Thrombosis or embolism events occurred within 6 months before enrollment;Anticoagulant therapy for therapeutic purposes (except low molecular weight heparin therapy) was used within 2 weeks prior to enrollment;Antiplatelet therapy is required.Current or recent (10 days before enrollment) use of aspirin (>325 mg/d), clopidogrel (>75 mg/d) or with dipyridamole, ticlopidine or cilostazol.Patients with metastatic lesions that invade the great vessels, respiratory tract, or mediastinum and are at significant risk of bleeding.

  10. underwent major surgery in the first 4 weeks of randomization, but did not include diagnostic biopsies.

  11. There have been CNS metastases 12. Severe unhealed wounds, active ulcers, and untreated fractures 13. Live vaccine was administered within 30 days prior to randomization. 14. An active autoimmune disease (i.e., immunoregulatory drugs, corticosteroids, or immunosuppressive drugs) requiring systemic treatment in the past 2 years;However, alternative therapy (such as thyroxine, insulin, or physiological corticosteroid replacement for adrenal or pituitary insufficiency) is not considered a systemic treatment and is permitted for use and inclusion.

  15. A history of definite interstitial lung disease or non-infectious pneumonia, unless caused by local radiotherapy;A history of active tuberculosis.

  16. Any severe acute or chronic infection requiring systemic antimicrobial, antifungal or antiviral treatment at the time of screening, excluding viral hepatitis.

  17. A history of human immunodeficiency virus (HIV) infection is known. 18. Previous allogeneic stem cell or solid organ transplantation. 19. Inability to swallow tablets, malabsorption syndrome, or any condition that affects gastrointestinal absorption.

  20. A history of severe allergy to any monoclonal antibody, anti-angiogenic target drug is known.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-05-11 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
PFS | 1.5 years
  Mainly observe the PFS of HCC patients
OS | 1.5 year
  Mainly observe the OS of HCC patients

CONTACTS AND LOCATIONS:
Locations (1):
- Fuda Cnacer Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided